CLINICAL TRIAL: NCT06801457
Title: Adjuvant Cerebroprotection Using Normobaric Hyperoxia in Pre-hospital Patients with Suspected Stroke
Acronym: AN-O2-EMS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AN-O2-EMS
Record Dates: First submitted 2025-01-21; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Stroke Acute
Keywords: Ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NBO (Experimental): NBO will be conducted with inhalation of 100% oxygen. NBO will be used in conjunction with best medical practice.
  Interventions: Other: NBO
- Control (Other): Best medical treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: NBO — NBO will be conducted with inhalation of 100% oxygen.
  Arms: NBO
Other: Control — Best medical care
  Arms: Control

SUMMARY:
The primary objective of this study is to determine the efficacy and safety of inhaled normobaric hyperoxia therapy (NBO) beginning in the pre-hospital setting in patients with suspected acute cerebral ischemia (ACI) due to large vessel occlusion presenting within 6 hours of symptom onset.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability globally, with acute ischemic stroke (AIS) patients often benefiting from intravenous thrombolysis and endovascular therapies such as mechanical thrombectomy, which have been shown to improve reperfusion rates. However, despite reperfusion, the proportion of patients with large vessel occlusion achieving a favorable functional outcome, defined as a modified Rankin Scale score of 0-2 at 90 days, remains under 50%.

Normobaric hyperoxia (NBO) emerges as a compelling option for cerebral protection. Its neuroprotective mechanisms are thought to include hypoxic tissue rescue, blood-brain barrier preservation, brain edema reduction, neuroinflammation alleviation, mitochondrial function improvement, oxidative stress mitigation, and apoptosis inhibition. NBO's diffusion properties allow it to reach the penumbra before reperfusion, enhancing aerobic metabolism and potentially reducing infarct volume. Its advantages also include low cost, wide availability, and ease of use, making it accessible across various healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old;
* Signs and symptoms are consistent with a new acute stroke, with low possibility of stroke mimics (e.g., no sudden coma, prior seizure disorder, suspected hypoglycemia);
* No prior stroke;
* The time from stroke onset/last seen well to randomization is within 6 hours;
* Paramedic-obtained FAST-ED score >= 3 (The enrollment of patients with a FAST-ED score of 3 is prespecified to constitute no more than 10% of the total study population);
* No significant pre-stroke disability (pre-stroke mRS 0-1);
* Signed informed consent from the patient or the legally authorized representative (LAR).

Exclusion Criteria:

* Endotracheal intubation in the field (prior to consent);
* Respiratory rate <= 10 or >= 30 breaths per minute;
* Oxygen-dependence at baseline to maintain SaO2 > 95%;
* Known history of severe chronic obstructive pulmonary disease (FEV1 less than 1.0), New York Heart Association (NYHA) Heart Failure Class III, acute pulmonary infection or aspiration pneumonia, prior to enrollment;
* Seizure at stroke onset;
* Exhibiting symptoms of vomiting, severe headache, or unconscious;
* Known pregnancy: women of childbearing age (18 to 44 years old according to the CDC's Division of Reproductive Health) will be asked about their pregnancy status.
* Participating in another clinical trial, or completed participation within prior 30 days;
* Receiving other neuroprotective agent (e.g., edaravone dexborneol, n-butylphthalide);
* Life expectancy < 90 days due to comorbidities;
* Unlikely to complete the 90-day follow-up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Level of disability at 90 days measured by modified Rankin scale (mRS) score | 90 days after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome; the primary outcome here is 3-month ordinal mRS score with mRS 5 and 6 merged into one category; modified intention-to-treat analysis

SECONDARY OUTCOMES:
Functional independence at 90 days defined as the proportion of patients with a modified Rankin scale (mRS) score of 0-2 at 90-day follow up | 90 days after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome. The mRS score is dichotomized to define the functional independence as mRS score of 0-2.
Excellent functional outcome at 90 days, defined as the proportion of patients with a modified Rankin scale (mRS) score of 0-1 at 90-day follow up | 90 days after randomization
  The original modified Rankin scale (mRS) ranges from 0 to 6, with higher scores indicating a worse outcome. The mRS score is dichotomized to define the excellent functional outcome as mRS score of 0-1.
National Institutes of Health Stroke Scale (NIHSS) obtained obtained upon Endovascular Thrombectomy (EVT) site arrival | Day 0
  The National Institutes of Health Stroke Scale (NIHSS) ranges from 0 to 42 points, with higher scores indicating worse neurological deficits. This is obtained upon Endovascular Thrombectomy (EVT) site arrival.
National Institutes of Health Stroke Scale (NIHSS) obtained at 24 hours | 24 hours after randomization
  The National Institutes of Health Stroke Scale (NIHSS) ranges from 0 to 42 points, with higher scores indicating worse neurological deficits.
ASPECTS on admission head CT | Day 0
  Alberta Stroke Program Early CT (ASPECT) score ranges from 0 to 10, with 10 being normal and 0 indicating complete MCA infarction obtained upon Endovascular Thrombectomy (EVT) site arrival.
NCCT infarct volume at 24 hours in patients undergoing thrombolysis or EVT (standard of care) | 24 hours after randomization
  Infarct volume measured by NCCT
Proportion of patients with elevated troponin level upon EVT hospital arrival | Day 0
  0-100%. This measure is obtained upon Endovascular Thrombectomy (EVT) site arrival.

OTHER OUTCOMES:
Serious adverse events/Adverse events | Through study completion
  total number of serious adverse events/adverse events reported during follow-up, according to standard definitions
Symptomatic intracranial hemorrhage | Up to 36 hours after randomization
  Number of cases of symptomatic intracerebral hemorrhage according to standard definition
Any intracranial hemorrhage | Up to 36 hours after randomization
  Number of cases of any intracranial hemorrhage according to standard definitions
Early neurological deterioration | 24 hours after randomization
  Early neurological deterioration at 24 hours, defined as at least 4-point increase in National Institutes of Health Stroke Scale (NIHSS) score from baseline; Larger the increase means worsening of outcomes. The Increase of score range from 0 to 42.
Heart rate at the end of oxygen therapy | Day 0
  Vital signs at the end of oxygen therapy
Respiratory rate at the end of oxygen therapy | Day 0
  Vital signs at the end of oxygen therapy
Systolic blood pressure at the end of oxygen therapy | Day 0
  Vital signs at the end of oxygen therapy
Diastolic blood pressure at the end of oxygen therapy | Day 0
  Vital signs at the end of oxygen therapy
Oxygen saturation at the end of oxygen therapy | Day 0
  Vital signs at the end of oxygen therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided